CLINICAL TRIAL: NCT04469114
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-design Trial of Tofacitinib in Hospitalized Participants With COVID-19 Pneumonia
Brief Title: Tofacitinib in Hospitalized Patients With COVID-19 Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 34810620.0.1001.0071
Record Dates: First submitted 2020-07-10; First posted 2020-07-13 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2020-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tofacitinib (Experimental): Tofacitinib 10mg twice daily for 14 days or until hospital discharge
  Interventions: Drug: Tofacitinib 10 mg
- Placebo (Placebo Comparator): Placebo twice daily for 14 days or until hospital discharge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tofacitinib 10 mg — Tofacitinib 10mg administered orally twice daily for 14 days or until hospital discharge
  Arms: Tofacitinib
Drug: Placebo — Tofacitinib-matching placebo administered orally twice daily for 14 days or until hospital discharge
  Arms: Placebo

SUMMARY:
Tofacitinib suppresses pro-inflammatory signaling that may be important pathogenetically to progression to more severe lung disease and acute respiratory distress syndrome (ARDS) in patients with COVID-19. The purpose of the study is to assess the safety and efficacy of tofacitinib plus standard pharmacologic and supportive measures in treating hospitalized participants with COVID-19 pneumonia.

DETAILED DESCRIPTION:
COVID-19 is a viral disease caused by a novel coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), that can cause severe pneumonia and ARDS. Respiratory viral load may peak within 5 days after onset, while symptoms are still mild. Many patients rapidly (within 1 to 2 weeks of infection) develop dyspnea and pneumonia and require hospitalization for respiratory support.

Preliminary clinical data from COVID-19 patients indicate that severe symptoms with SARS-CoV-2 infection are associated with an exaggerated immune response driven by interleukin (IL)-6 IL-10, tumor necrosis factor (TNF)α, and other cytokines. The ultimate result is progressive destruction of the alveolar epithelium leading to pneumonia and/or ARDS. Moreover, the exudative phase of ARDS is thought to be due to an influx of myeloid cells (neutrophils and macrophages) and elevations of inflammatory cytokines, with higher levels of both IL-6 and IL-8 levels being correlated with increased mortality. Therefore, immunomodulatory therapy may be beneficial in reducing the deleterious effects of lung inflammation and mitigating progressive lung injury.

Tofacitinib is an inhibitor of Janus kinase (JAKs) 1 and 3, with partial selectivity to JAK 2. Tofacitinib suppresses pro-inflammatory signaling that may be important pathogenetically to progression to more severe lung disease and ARDS in patients with COVID-19.

The purpose of the study is to assess the safety and efficacy of tofacitinib plus standard pharmacologic and supportive measures in treating hospitalized participants with COVID-19 pneumonia.

Participants with laboratory confirmed SARS-CoV-2 infection as determined by a positive PCR, who have agreed to participate, will be screened within 72h hours after admission to the hospital to determine eligibility.

Eligible participants will be randomized on Day 1 to the tofacitinib plus standard of care treatment group or the placebo plus standard of care treatment group in a 1:1 ratio, stratified by site. Participants will receive treatment for up to 14 days or until discharge from the hospital, whichever is earlier.

Participants will be assessed daily (up to Day 28) while hospitalized for clinical, safety, and laboratory parameters. Follow-up visits will occur on Day 14 and on Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants older than 18 years
2. Laboratory-confirmed novel coronavirus (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR) prior to Day 1.
3. Evidence of pneumonia assessed by radiographic imaging (chest x-ray or chest CT scan).
4. Hospitalized for less than 72 hours and receiving supportive care for COVID-19

Exclusion Criteria:

1. Require non-invasive ventilation, invasive mechanical ventilation, or extracorporeal membrane oxygenation (ECMO) on Day 1 at the time of randomization
2. History of or known current thrombosis. Only if current thrombosis is suspected by the investigator, imaging testing is recommended (per local guidance) to exclude thrombosis.
3. Have a personal or first-degree family history of blood clotting disorders.
4. Participants who are immunocompromised, with known immunodeficiencies, or taking potent immunosuppressive agents (eg, azathioprine, cyclosporine).
5. Participants with any current malignancy or lymphoproliferative disorders that requires active treatment
6. Severe hepatic impairment, defined as Child-Pugh class C.
7. Severe anemia (hemoglobin <8 g/dL).
8. Absolute lymphocyte count <500 cells/mm;
9. Absolute neutrophil count <1000 cells/mm.
10. Known allergy to tofacitinib.
11. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk associated with study participation or, in the investigator's judgment, make the participant inappropriate for the study.
12. Suspected or known active systemic bacterial, fungal, or viral infections (with the exception of COVID-19) including but not limited to: active herpes zoster infection; known active tuberculosis or history of inadequately treated tuberculosis; known B hepatitis, C hepatitis, or HIV.
13. Have received any of these within 4 weeks prior to the first dose of study intervention: any JAK inhibitors, potent immunosuppressants, or any biologic agents including IL-6 inhibitors (eg, tocilizumab) or IL-1 inhibitors (eg, anakinra) within the past 30 days; any potent cytochrome P450 inducer, such as rifampin, within the past 28 days or 5 half-lives, whichever is longer.
14. Have received estrogen-containing contraception or treatment with herbal supplements within 48 hours prior to the first dose of study intervention.
15. Have received treatment with corticosteroids equivalent to prednisone or methylprednisolone >20 mg/day for equal or more than 14 consecutive days prior to screening.
16. Current participation in other trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Death or respiratory failure until Day 28 | 28 days
  1, 2 or 3 on the 8-point National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale of disease severity. The minimum value is 1 (worst outcome) and the maximum value is 8 (best outcome).
  1. Death.
  2. Hospitalized, on invasive mechanical ventilation or ECMO.
  3. Hospitalized, on non-invasive ventilation or high-flow oxygen devices.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise).
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care.
  7. Not hospitalized, limitation on activities and/or requiring home oxygen.
  8. Not hospitalized, with no limitations on activities.

SECONDARY OUTCOMES:
National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale of disease severity at Day 14 | 14 days
  NIAID ordinal scale of disease severity
Status of alive and not on mechanical ventilation or ECMO at Day 14 and 28 NIAID ordinal scale of disease severity at Day 14 | 14 and 28 days
  Categories 3 to 8 in the National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale of disease severity at Day 14 and Day 28
Status of requiring supplemental oxygen at Day 28 | 28 days
  Categories 1 to 4 in the National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale of disease severity
Status of being alive and not hospitalized at Day 14 and 28 | 14 and 28 days
  Categories 7 and 8 in the National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale of disease severity
National Institute of Allergy and Infectious Diseases (NIAID) ordinal scale of disease severity at Day 14 NIAID ordinal scale of disease severity at Day 28 | 28 days
  NIAID ordinal scale of disease severity
Number of patients with cure | 28 days
  Number of patients with resolution of fever, cough, and need for ventilatory or oxygen support.
Number of patients at the ICU or on ventilatory support at Day 28 | 28 days
  Number of patients at the ICU or on ventilatory support
Number of days free from mechanical ventilation at 28 days | 28 days
  Number of days free from mechanical ventilation
Number of days in hospital | 28 days
  Number of days in hospital
Number of days in ICU | 28 days
  Number of days in ICU
Death or respiratory failure at Day 28 | 28 days
  Categories 1 to 3 in the National Institute of Allergy and Infectious Diseases (NIAID)

CONTACTS AND LOCATIONS:
Locations (17):
- Brazil (17):
  - Centro de Pesquisa Clínica do Coração, Aracaju
  - Hospital Universitário São Francisco de Assis Na Providência de Deu, Bragança Paulista
  - Irmandade do Sr. Bom Jesus dos Passos da Santa Casa de Misericórdia de Bragança Paulista, Bragança Paulista
  - Hospital do Coração do Brasil, Brasília
  - Instituto de Pesquisa Clínica de Campinas, Campinas
  - Hospital Regional do Litoral Norte, Caraguatatuba
  - Unimed Fortaleza Sociedade Corporativa Médica LTD, Fortaleza
  - Hospital Regional Jorge Rossmann, Itanhaém
  - Hospital Bruno Born, Lajeado
  - Hospital São Vicente de Paulo, Passo Fundo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - Hospital Regional de Registro, São José dos Campos
  - Hospital Regional de São José dos Campos, São José dos Campos
  - Beneficência Portuguesa, São Paulo
  - BP Mirante, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Instituto do Coração, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guimaraes PO, Damiani LP, Tavares CAM, Halpern ASR, Deuring JJ, Rizzo LV, Berwanger O. Laboratory profiles of patients hospitalized with COVID-19 pneumonia treated with tofacitinib or placebo: a post hoc analysis from the STOP-COVID trial. Einstein (Sao Paulo). 2024 Nov 4;22:eAO0821. doi: 10.31744/einstein_journal/2024AO0821. eCollection 2024. PMID 39504090
- [Derived] Kramer A, Prinz C, Fichtner F, Fischer AL, Thieme V, Grundeis F, Spagl M, Seeber C, Piechotta V, Metzendorf MI, Golinski M, Moerer O, Stephani C, Mikolajewska A, Kluge S, Stegemann M, Laudi S, Skoetz N. Janus kinase inhibitors for the treatment of COVID-19. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD015209. doi: 10.1002/14651858.CD015209. PMID 35695334
- [Derived] Guimaraes PO, Quirk D, Furtado RH, Maia LN, Saraiva JF, Antunes MO, Kalil Filho R, Junior VM, Soeiro AM, Tognon AP, Veiga VC, Martins PA, Moia DDF, Sampaio BS, Assis SRL, Soares RVP, Piano LPA, Castilho K, Momesso RGRAP, Monfardini F, Guimaraes HP, Ponce de Leon D, Dulcine M, Pinheiro MRT, Gunay LM, Deuring JJ, Rizzo LV, Koncz T, Berwanger O; STOP-COVID Trial Investigators. Tofacitinib in Patients Hospitalized with Covid-19 Pneumonia. N Engl J Med. 2021 Jul 29;385(5):406-415. doi: 10.1056/NEJMoa2101643. Epub 2021 Jun 16. PMID 34133856